CLINICAL TRIAL: NCT02335671
Title: Evaluating Mass Spectrometry And Intraoperative MRI In The Advanced Multimodality Image Guided Operating Suite (Amigo) In Breast-Conserving Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Thanh Barbie, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 14-476
Record Dates: First submitted 2015-01-07; First posted 2015-01-12 (Estimated); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Early Stage Breast Cancer; Breast Cancer Stage I; Breast Cancer Stage II
Keywords: Early Stage Breast Cancer; Breast Conserving Surgery; Breast Cancer Stage I; Breast Cancer Stage II
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intra-operative Magnetic Resonance Imaging (MRI) (Experimental): * Preoperative diagnostic MRI
  * Intra-operative MRI
  * Standard lumpectomy and sentinel node biopsy if indicated, or standard axillary dissection if clinically indicated
  * Specimen to Pathology and Mass Spectrometer (Analysis of Tissue Sample)
  Interventions: Procedure: Intra-operative Magnetic Resonance Imaging (MRI); Other: Mass Spectrometer Analysis of Tissue Sample

INTERVENTIONS:
Procedure: Intra-operative Magnetic Resonance Imaging (MRI)
Other: Mass Spectrometer Analysis of Tissue Sample — Analysis of Tissue Sample

SUMMARY:
The purpose of this study is to investigate the use of intra-operative Magnetic Resonance Imaging (MRI) and Mass Spectrometry (MS) during breast conserving surgery, and to determine if these tests are capable of accurately predicting the presence or absence of breast tumor in surgical specimens at the margins.

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial investigating the use of intra-operative MRI and MS in breast cancer surgery. Phase II clinical trials test the safety and effectiveness of an investigational intervention to learn whether the intervention works in treating a specific disease. "Investigational" means that the intervention is being studied.

Prior research has shown that intraoperative MRI and MS are two types of tests that are feasible to use during cancer surgery and may be able to guide therapy. In this study, we are evaluating the accuracy of intra-operative MRI and MS in determining whether or not all cancer tissue was removed during breast surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be female
* Participants must have a pre-operative standard mammogram with or without ultrasound. These may be performed at outside institutions.
* Participants must have biopsy confirmed and clinical stage 1 or stage 2 breast carcinoma. If biopsy was done at an outside hospital, pathology will be reviewed at BWH/DFCI.
* Participants must be candidates for definitive local therapy with breast conserving therapy (this takes into account tumor to breast size ratio appropriate for BCS, and the ability to undergo standard radiation therapy post-operatively).
* Patient must meet standard MRI guidelines and be able and willing to undergo MRI
* Age ≥18 years and < 75.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Participants with a known BRCA 1 or 2 mutation.
* Participants with known Li-Fraumeni or Cowden's Disease.
* Participants with prior mantle radiation.
* Participants with locally advanced breast cancer such as inflammatory breast cancer or cancer grossly involving skin.
* Participants who are pregnant.
* Participants who enroll in a preoperative therapy trial or who have been treated with neoadjuvant chemotherapy.
* Participants with known active collagen vascular disease.
* Participants with prior history of ipsilateral breast carcinoma.
* Patients who have biopsy confirmed multi-centric disease.
* Participants who have documented contra-indications for contrast-enhanced MRI, including but not limited to renal failure.
* Participants who exceed the weight limit for the surgical table at AMIGO, 350 lbs or who will not fit into the 70 cm diameter bore of the MRI scanner at AMIGO or the 60 cm diameter bore of the pre-procedure imaging MRI scanner.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-02; Primary Completion 2023-01 (Actual); Study Completion 2023-01 (Actual)

PRIMARY OUTCOMES:
To evaluate the accuracy of MRI in detecting tumor boundaries | 2 Years

SECONDARY OUTCOMES:
To determine the operating characteristics (sensitivity, specificity, negative predictive value and positive predictive value) of MRI in detecting tumor boundaries as confirmed with pathologic results | 2 Years
To evaluate the correlation of intraoperative mass spectrometry results to tumor boundaries as confirmed with pathologic results. | 2 Years
To develop novel image processing algorithms to detect remnant tumor from intraoperative DCE-MRI in presence of tissue edema and reduced perfusion | 2 Years

CONTACTS AND LOCATIONS:
Overall Officials: Thanh Barbie, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts